CLINICAL TRIAL: NCT03545503
Title: A Randomized Controlled Trial to Evaluate the Hemodynamic Effects of Ketamine Versus Etomidate During Rapid Sequence Intubation
Brief Title: Evaluating the Hemodynamic Effects of Ketamine Versus Etomidate During Rapid Sequence Intubation
Acronym: Ket-RSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: South East Area Health Education Center, Wilmington, NC (Other)
Collaborators: New Hanover Regional Medical Center (Other)
Responsible Party: Principal Investigator, William F Powers, IV, MD, Assistant Professor of Surgery, South East Area Health Education Center, Wilmington, NC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1712-4
Record Dates: First submitted 2018-01-31; First posted 2018-06-04 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Intubation Complication
Keywords: Rapid Sequence Intubation; Hemodynamics; Etomidate; Ketamine
MeSH Terms: interventions — Etomidate; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etomidate (Active Comparator): Etomidate will be dosed once at a standard of 0.3 mg/kg via IV Push
  Interventions: Drug: Etomidate
- Ketamine (Active Comparator): Ketamine will be dosed once at a standard 2 mg/kg via IV Push
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Etomidate — Etomidate will be administered as the sedative for RSI on even days
  Other Names: Amidate
  Arms: Etomidate
Drug: Ketamine — Ketamine will be administered as the sedative for RSI on odd days
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
The purpose of this study is to compare the hemodynamic effects of ketamine v etomidate during rapid sequence intubation (RSI) in the pre-hospital and emergency department setting.

DETAILED DESCRIPTION:
This is a randomized prospective study evaluating the hemodynamic response in adult participants greater than or equal to 18 years of age undergoing RSI in the pre-hospital or emergency department setting. Hemodynamic response is the cardiology response of the circulatory system. The investigators will compare the drugs Ketamine and Etomidate in participants having RSI. Ketamine and Etomidate are immediately available for RSI in both settings as both are currently standards of care for RSI.

Research thus far demonstrates that both Etomidate and ketamine are safe and effective for RSI. Despite the reported safety of Ketamine, Etomidate usage continues to far surpass that of ketamine. Both Etomidate and Ketamine are FDA-approved for induction of anesthesia. They are both ideal drugs for intubation due to their pharmacokinetic properties including a quick onset of less than 60 seconds, a short duration of about 10 minutes, and the minimal effect they have on the cardiovascular system. The neutral effect on the cardiovascular system is particularly important in the acute and traumatic setting when patients are often hypotensive.

However, there are some differences and disadvantages in the two medications. Due to these factors and limited data to support Ketamine as an equal or superior alternative to Etomidate, it has been difficult to clearly recommend one agent over the other for RSI.

Data will be analyzed using SPSS with a p-value of less than 0.05 being considered significant. The PI will consider a 20% decrease in systolic BP from a participant baseline as significant, and will compare the incidence of post RSI hypotension between the two groups. Several a priori subgroups will be evaluated to include patients greater than 70 years of age, trauma participants requiring RSI, and those participants whose shock index is less than 0.9 versus those whose shock index is greater than 0.9.

To maintain 80% power with a probability of 0.05, 200 participants will be needed in each arm to detect at 25% difference in SBP (baseline to post drug administration effects)

ELIGIBILITY:
Inclusion Criteria:

* Persons greater than 18yrs requiring rapid sequence intubation for any reason.

Exclusion Criteria:

* Pregnant patients
* Children under the age of 18
* Patients with a known hypersensitivity to etomidate or ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F Powers IV, MD, Principal Investigator — New Hanover Regional Medical Center
Locations (1):
- New Hanover Regional Medical Center, Wilmington, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited if they required rapid sequence intubation in the pre-hospital or 17th street campus emergency department setting between January 1, 2018 and July 30, 2019.
Pre-assignment Details: 98 did not meet inclusion criteria, 48 had incomplete sedative data, and 71 were excluded for other reasons
Period: Overall Study
Arm/Group | Etomidate | Ketamine
Started | 208 | 220
Completed | 194 | 204
Not Completed | 14 | 16
Not completed — Protocol Violation | 14 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etomidate | Ketamine | Total
Number analyzed (Participants) | 194 | 204 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.48 (19.5) | 56.68 (19.68) | 57.08 (19.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 74 | 141
  Male | 127 | 130 | 257
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamic Effect as Measured by Systolic Blood Pressure Before and After RSI
Description: The primary outcome of this study is to determine the change in hemodynamic response comparing systolic blood pressure pre-versus post-administration of study drug. A significant hemodynamic response is defined as a decrease in systolic blood pressure of 20% or greater between the pre versus post administered study drug.
Time Frame: The hemodynamic response will be measured by assessing the change in vital signs between 15 minutes prior to administration and vitals up to 15 minutes after the administration of the study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Etomidate: Participants randomized to receive etomidate
- Ketamine: Participants randomized to receive ketamine
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 194 | 204
mmHg
  Pre-SBP | 138.04 (38.63) | 132.39 (39.54)
  Post SBP 0-7 | 139.09 (44.52) | 130.09 (41.78)
  Post SBP 8-15 | 130.42 (42.19) | 120.80 (37.37)

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Etomidate: Participants receiving etomidate
- Ketamine: Participants receiving ketamine
Arm/Group | Etomidate | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/204
Serious Adverse Events (participants affected / at risk) | 0/194 | 1/204
Other Adverse Events (participants affected / at risk) | 117/194 | 111/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etomidate (N=194) | Ketamine (N=204)
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etomidate (N=194) | Ketamine (N=204)
Hypertension (Vascular disorders) | 117 | 111 — AE for HTN grade 2 and 3 is being reported here regardless of the attribution.
Hypotension (Vascular disorders) | 36 | 53 — AE for hypotension is being reported regardless of the grade and attribution. Note: Gr 4 is challenging to capture as participants were already being hospitalized due to their underlying condition.

LIMITATIONS AND CAVEATS:
Investigators nor clinicians were blinded to study drug. Resuscitation pre-RSI was not accounted for nor was the dosing for vascopressors. We could not control the slow administration of ketamine to decrease effects of hypotension due to rapid administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03545503/Prot_SAP_000.pdf